CLINICAL TRIAL: NCT06733727
Title: A Randomized Double-blind Placebo-controlled Trial Comparing Letrozole Versus Mifepristone As Pre-treatment Before Medical Management of First Trimester Silent Miscarriage Using Misoprostol
Brief Title: Letrozole Versus Mifepristone and Misoprostol in Silent Miscarriage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Kwong Wah Hospital (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW22-530
Record Dates: First submitted 2024-12-06; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-08

CONDITIONS: Silent Miscarriage
Keywords: silent miscarriage; mifepristone; misoprostol; letrozole
MeSH Terms: conditions — Abortion, Incomplete | interventions — Letrozole; Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Active Comparator): Letrozole 10mg per day from day 1-3 orally, placebo mifepristone Sublingual misoprostol 800 microgram on day 3
  Interventions: Drug: Letrozole
- Mifepristone (Active Comparator): Mifepristone 200mg orally on day 1, placebo letrozole on day 1-3 Sublingual misoprostol 800 microgram on day 3
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Letrozole — Letrozole pre-treatment in addition to misoprostol as medical management for silent miscarriage
  Arms: Letrozole
Drug: Mifepristone — Mifepristone pre-treatment in addition to misoprostol as medical management for silent miscarriage
  Other Names: Mifepristone, RU486
  Arms: Mifepristone

SUMMARY:
Management of first trimester silent miscarriage can be by expectant, medical or surgical management. Surgical management by suction evacuation is associated with surgical risks (including risks to the womb that can affect further pregnancy), anaesthetic risks and hospital stay. Medical management of first trimester silent miscarriage using misoprostol is another common option that can reduce the risk of bleeding and those associated with surgery. However, the current standard management of using misoprostol for the management of first trimester miscarriage only has a success rate of 70-80%, which is suboptimal.

Recent large studies have shown that adding mifepristone pre-treatment before misoprostol in the management of silent miscarriage can improve the success rates of complete miscarriage after medical management. There are 2 problems with mifepristone. Firstly, it is not widely available in many countries for cultural and religious reasons because it is labelled as an 'abortifacient'. Secondly, it is expensive. One tablet of Mifepristone costs $500 HK dollars. There is a need to look for an alternative to mifepristone.

Letrozole is an aromatase inhibitor which can reduce estrogen levels. Some studies have shown that it can improve the success rate of medical management of silent miscarriage and termination of pregnancy. It is safe, more widely available and cheaper than mifepristone.

This is a randomized double blinded trial comparing the use of mifepristone versus letrozole as pre-treatment in the medical management of first trimester silent miscarriage using misoprostol.

DETAILED DESCRIPTION:
This is a randomized double blinded trial comparing the use of mifepristone versus letrozole as pre-treatment in the medical management of first trimester silent miscarriage using misoprostol.

Both groups will receive misoprostol (which is the standard management for medical management of silent miscarriage locally), but they will be randomized to either adding mifepristone or letrozole as pre-treatment. Mifepristone is usually taken once 2 days before misoprostol, whereas letrozole is taken 10mg daily for 3 days before misoprostol. Placebo of letrozole and mifepristone will be given to maintain double blindness of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with silent miscarriage <= 12 weeks of gestation by ultrasonography
* Single intrauterine gestational sac
* No heavy per-vaginal bleeding
* No severe abdominal pain
* No features of intrauterine infection
* Able to understand the proposed research and able to comply with instructions
* Having given voluntary written informed consent

Exclusion Criteria:

* Known allergy to mifepristone, misoprostol or letrozole
* On drugs with potential drug interactions with mifepristone e.g. aspirin, clopidogrel, anti-coagulants etc.
* Suspected ectopic or molar pregnancy or multiple pregnancy
* Distorted uterine cavity by uterine septum or submucosal fibroids
* Presence of intrauterine contraceptive device
* History of bleeding tendencies e.g. haemorrhagic diseases, current anti-coagulant treatment
* Previous history of retained products of gestation/ failed medical management of miscarriage
* Opt for expectant or surgical management of miscarriage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 884 (Estimated)
Dates: Start 2024-12-06 (Estimated); Primary Completion 2027-12-05 (Estimated); Study Completion 2028-06-05 (Estimated)

PRIMARY OUTCOMES:
Gestational sac expulsion | 2 weeks, 30 days
  Gestational sac expulsion by the first follow up visit after 2 weeks of misoprostol administration and no additional surgical or medical intervention within 30 days after randomization

SECONDARY OUTCOMES:
Time of tissue expulsion | 6 weeks
  Time of tissue expulsion
Return of normal menses | 6 weeks
  Return of normal menses without additional intervention
Requirement of repeated intervention | 6 weeks
  Requirement of repeated intervention including repeated course of medical treatment or surgery
Unplanned re-admission | 6 weeks
  Number of unplanned re-admission
Analgesics | 6 weeks
  Use of analgesics
Side effects | 6 weeks
  Vomiting
Side effects | 6 weeks
  Nausea
Side effects | 6 weeks
  Fever
Side effects | 6 weeks
  Diarrhoea
Side effects | 6 weeks
  Abdominal pain on a visual analog scale
Vaginal bleeding | 6 weeks
  Duration and amount of vaginal bleeding
Complications | 6 weeks
  Including severe vaginal bleeding requiring transfusion, infection
Return of menstruation | 6 weeks
  Timing of return of menses
Women's satisfaction | 6 weeks
  Client satisfaction questionnaire
Women's satisfaction | 6 weeks
  EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ko, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan at the current moment